CLINICAL TRIAL: NCT01185912
Title: Cardiomyocyte Apoptosis Following Antegrade and Retrograde Cardioplegia
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Finnish Foundation for Cardiovascular Research (Other)
Responsible Party: Principal Investigator, Markus Malmberg, MD, Turku University Hospital
Other Study IDs: 1/2006
Record Dates: First submitted 2010-06-24; First posted 2010-08-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Cardiomyocyte Apoptosis
Keywords: Cardiac MRI; Cardiac ultrasound; Cardiac surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Transmyocardial needle biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiomyocyte apoptosis: Elective aortic valve replacement patience
  Interventions: Procedure: Ventricle muscle tissue samples

INTERVENTIONS:
Procedure: Ventricle muscle tissue samples

SUMMARY:
Retrograde cardioplegia during heart surgery is associated with inadequate myocardial protection. In experimental animal study retrograde cardioplegia induces more cardiomyocyte apoptosis when compared to antegrade cardioplegia. 20 volunteer patients under going elective aortic valve surgery will be divided in to two groups: 10 patients receiving only antegrade cardioplegia and 10 patients receiving only retrograde cardioplegia. Pre- and post-operatively cardiac MRI and cardiac ultrasound will be performed. During the surgery ventricular muscle samples will be taken in order to assess cardiomyocyte apoptosis. Aims of the study: 1. whether the cardiomyocyte apoptosis is significantly more induced after retrograde cardioplegia than antegrade cardioplegia, 2. whether the amount of apoptotic cardiomyocytes correlates to conventional markers of myocardial injury after cardiac surgery, 3. whether the extent of irreversible myocardial damage by apoptosis correlates to post-ischemic contractile dysfunction after cardiac surgery, as measured with echocardiography, 4. whether the amount of cardiomyocyte apoptosis correlates to long term outcome and cardiac function as measured with MRI.

ELIGIBILITY:
Inclusion Criteria:

* aortic valve stenosis or combined aortic valve disease

Exclusion Criteria:

* angiographically verified hemodynamically significant coronary artery disease impaired left ventricular function (left ventricular ejection fraction <50%) surgery including additional procedures other than aortic valve replacement cancer

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients (male and female) undergoing elective aortic valve replacement surgery due to aortic valve stenosis or combined aortic valve disease in Turku University Hospital, Department of Surgery.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Department of Surgery, Turku, Finland